CLINICAL TRIAL: NCT03592589
Title: Prevention of Atelectasis, Via High Flow Nasal Cannula to Obtain a PEP, During General Anesthesia for MRI by Sevoflurane in Children, Evaluated by Lung MRI and Echography
Brief Title: Prevention of Atelectasis, Via High Flow Nasal Cannula to Obtain a PEP, During General Anesthesia in Children
Acronym: PREVAT-PED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-39
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): standard general anesthesia using sevoflurane delivered by a pediatric high concentration mask
- Intervention group (Experimental): sevoflurane will be deliver by a pediatric high flow nasal canula (2L/KG/min)
  Interventions: Device: high flow nasal canula

INTERVENTIONS:
Device: high flow nasal canula — high flow nasal canula to obtain a positive expiratory pressure
  Arms: Intervention group

SUMMARY:
Anesthesia causes respiratory changes and complications, which are the main causes of complications and anesthesia-related deaths.

Among the complications, the rapid appearance of lung atelectasis is well known, deteriorating the hematosis during anesthesia, and inducing secondary pulmonary complications.

Prevention or limitation of the atelectasis would be a way to improve the safety of patients who have a limited respiratory function.

The application of a positive expiratory pressure (PEP) is an effective prevention method for atelectasis, that have been only demonstrate in patients under mechanical ventilation.

The high flow nasal cannula is a non-invasive technique easy to perform and allowing a PEP. High flow nasal cannula is safe to use, and the interface is free from local skin complications.

Chest X-ray (bad sensibility) or CT are usually used for the diagnosis of atelectasis, but these two exams involve irradiation for patient. MRI and pulmonary ultrasonography has now been validated in adults. MRI are relatively long, and allow to investigate the atelectasis with only a short additional acquisition time.

Thus, it would be the first study on the effect of the PEP on the impact and the volume of the atelectasis during general anesthesia in spontaneous ventilation in children. By the way this is the first study on lung's anatomical effects of high flow nasal cannula.

It is a monocentric, intervention, randomized, superiority study whose main purpose is to show the reduction of the atelectasis through the use of high flow nasal cannula versus a high concentration mask for pediatric anesthesia during MRI.

The studied population is all the children between 6 months and 5 years with a pediatric indication of general anesthesia for MRI.

The primary goal is to show a reduction of volume (cm3) of the atelectasis via the application of a PEP by high flow nasal cannula.

The main assessment criteria is the ratio of atelectasis volume/total lung volume.

The prevalence of the atelectasis will be evaluated by MRI lung and measured using 3D reconstruction software. The duration of the examination and the anesthesia is slighty lengthened, 3 to 5 minutes for a 40 minutes' exam.

The secondary objective is to show a match between the atelectasis on MRI and ultrasound.

DETAILED DESCRIPTION:
Anesthesia causes respiratory changes and complications, which are the main causes of complications and anesthesia-related deaths.

Among the complications, the rapid appearance of lung atelectasis is well known, deteriorating the hematosis during anesthesia, and inducing secondary pulmonary complications.

Prevention or limitation of the atelectasis would be a way to improve the safety of patients who have a limited respiratory function.

The application of a positive expiratory pressure (PEP) is an effective prevention method for atelectasis, that has been demonstrated only in patients under mechanical ventilation.

The high flow nasal cannula is a non-invasive technique easy to perform and allowing a PEP. High flow nasal cannula is safe to use, and the interface is free from local skin complications.

Chest X-ray (bad sensibility) or CT are usually used for the diagnosis of atelectasis, but these two exams involve irradiation for patient. MRI and pulmonary ultrasonography has now been validated in adults. The investigators has a long experience of anesthesia in spontaneous ventilation in children for MRI. MRI are relatively long, and allow to investigate the atelectasis with only a short additional acquisition time.

Thus, it would be the first study on the effect of the PEP on the impact and the volume of the atelectasis during general anesthesia in spontaneous ventilation in children. By the way this is the first study on lung's anatomical effects of high flow nasal cannula.

It is a monocentric, intervention, randomized, superiority study whose main purpose is to show the reduction of the atelectasis through the use of high flow nasal cannula versus a high concentration mask for pediatric anesthesia during MRI.

The studied population is all the children between 6 months and 5 years with a pediatric indication of general anesthesia for MRI.

The primary goal is to show a reduction of volume (cm3) of the atelectasis via the application of a PEP by high flow nasal cannula.

The main assessment criteria is the ratio of atelectasis volume/total lung volume.

The prevalence of the atelectasis will be evaluated by MRI lung and measured using 3D reconstruction software. The duration of the examination and the anesthesia is slighty lengthened, 3 to 5 minutes for a 40 minutes' exam.

The secondary objective is to show a match between the atelectasis on MRI and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Indication of general anesthesia for MRI
* Patient between 6 months and 5 years old
* ASA score I or II
* No facial dysmorphia
* No predicting difficult intubation
* Parental consent

Exclusion Criteria:

* Severe cardio-pulmonary disease
* Lack of coverage by health insurance
* ASA III or IV
* Parental refuse for inclusion

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
atelectasis volume by Lung MRI | 40 minutes
  volume (cm3) of the total lung.
  The main assessment criteria is the ratio of atelectasis volume/total lung volume.
  The prevalence of the atelectasis will be evaluated by MRI lung and measured using 3D reconstruction software.
total lung volume by Lung MRI | 40 minutes
  volume (cm3) of the atelectasis via the application of a PEP by high flow nasal cannula.
  The main assessment criteria is the ratio of atelectasis volume/total lung volume.
  The prevalence of the atelectasis will be evaluated by MRI lung and measured using 3D reconstruction software.

SECONDARY OUTCOMES:
atelectasis volume by lung ultrasonography | 15 to 45 minutes after begining general anesthesia
  Lung ultrasonography will be pratice in recovery room, just after the MRI. The Lung ultrasonography score will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Roncin C, Scemama U, Zieleskiewicz L, Loundou A, Lesavre N, Vialet R. Atelectasis prevention during anaesthesia using high-flow nasal cannula therapy: A paediatric randomised trial using MRI images. Anaesth Crit Care Pain Med. 2020 Dec;39(6):819-824. doi: 10.1016/j.accpm.2020.08.009. Epub 2020 Oct 17. PMID 33080406